CLINICAL TRIAL: NCT06729671
Title: A Probiotic Strategy for Antipsychotic-induced Metabolic Dysfunction
Acronym: MetaboMicrobe
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College Cork (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: APC175
Record Dates: First submitted 2024-11-19; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Psychosis
Keywords: microbiota; antipsychotic; weight gain
MeSH Terms: conditions — Psychotic Disorders; Weight Gain | interventions — Capsules; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placebo (Placebo Comparator): hydroxypropylmethylcellulose (HPMC) capsule with maltidextrin
  Interventions: Dietary Supplement: maltodextrin
- active (Active Comparator): Bifidobacterium longum APC1472 hydroxypropylmethylcellulose (HPMC) capsules
  Interventions: Dietary Supplement: Bifidobacterium longum APC1472 hydroxypropylmethylcellulose (HPMC) capsule

INTERVENTIONS:
Dietary Supplement: Bifidobacterium longum APC1472 hydroxypropylmethylcellulose (HPMC) capsule — Bifidobacterium longum APC1472 capsule
  Arms: active
Dietary Supplement: maltodextrin — maltodextrin
  Arms: placebo

SUMMARY:
Antipsychotic drugs are used to treat a range of psychiatric disorders including schizophrenia, bipolar disorders, and psychotic depression. Most antipsychotics are associated with significant weight gain and metabolic disturbances, which increase the risks for other diseases (obesity, diabetes, coronary diseases, etc.) and negatively impact medication adherence and quality of life. Evidence has shown that Olanzapine, for example, increases appetite, food intake, and food reward and modulates the gut microbiota. The gut microbiota can modulate adiposity, metabolism and immune-endocrine signals that impact host's energy balance and feeding behaviour. This, together with the fact that antipsychotic-induced remodelling of the gut microbiota has been associated with weight gain, suggests that microbiota-targeted interventions could help to alleviate or prevent the distressing side-effects of antipsychotic medications. The investigators have previously published promising data demonstrating anti-obesity effects of a novel Bifidobacterium longum APC1472, in a mouse model of obesity and in an overweight/obese population of humans, reducing levels of glucose and normalizing ghrelin levels. Because atypical antipsychotic medications are often used in people experiencing psychosis and the mechanisms of antipsychotic-induced weight gain and metabolic dysfunction have been suggested to include glucose intolerance (hyperglycaemia) and aberrant ghrelin signalling, the investigators propose to assess if adjunct supplementation of Bifidobacterium longum APC1472 can attenuate weight gain and metabolic side-effects associated with the use of atypical antipsychotic medication in people with non- affective psychosis. The investigators propose an exploratory patient-oriented research study, to assess the potential of adjunct Bifidobacterium longum APC1472 supplementation in individuals with psychosis receiving antipsychotic treatment, to ameliorate the liability to gain weight and/or normalize metabolic disturbances. Findings from this study will support clinical decision-making, increasing patient choice, and increase medication adherence, which will ultimately improve health and quality of life, and overall wellbeing of individuals as they pass through normal life stages.

DETAILED DESCRIPTION:
Schizophrenia is a mental illness associated with psychosis and is treated with antipsychotic medication. These medications are very effective; however, they are associated with side-effects that impact people's physical health. Substantial body weight gain occurs in up to half of people during long-term antipsychotic treatment. Antipsychotics can also increase glucose (sugar) and lipid (fat) levels in the blood, and the ones that do this the most, tend to be the same ones that cause the most weight gain. People taking antipsychotics regard weight gain as one of the most distressing side-effects caused by their medication. This weight gain often leads people to stop taking their antipsychotic treatment with a risk of their psychosis returning. People with psychosis die 15-20 years earlier than the general population. The leading cause of 'years of life' lost in this population is poor physical health. Heart disease and metabolic disorders are 1.4-2-fold more common in this population. Being overweight increases the risk of heart attack, stroke, and developing many physical illnesses and cancers. Furthermore, being overweight and experiencing psychosis are associated with reduced self-esteem, reduced quality of life, and stigma.

In a previous study by the investigating team, the investigators found that a bacteria found in the gut of healthy individuals, Bifidobacterium longum APC1472, was able to prevent obesity in mice treated with an antipsychotic. A second study conducted by the investigating team with people who were overweight or obese found that this type of bacteria, which may be developed into a new probiotic, improved sugar levels. The investigators are now looking to examine the impact this bacteria could have on the weight, blood sugars, and wellbeing of people treated with antipsychotic medication. Having access to a probiotic capsule that alleviates the most distressing side-effects of antipsychotic medications will benefit people who need these medications greatly.

Antipsychotic drugs are used to treat a range of psychiatric disorders including schizophrenia, bipolar disorders, and psychotic depression. Most antipsychotics are associated with significant weight gain and metabolic disturbances, which increase the risks for other diseases (obesity, diabetes, coronary diseases, etc.) and negatively impact medication adherence and quality of life. Evidence has shown that olanzapine, for example, increases appetite, food intake, and food reward and modulates the gut microbiota. The gut microbiota can modulate adiposity, metabolism and immune-endocrine signals that impact host's energy balance and feeding behaviour. This, together with the fact that antipsychotics induced remodeling of the gut microbiota has been associated with weight gain, suggests that microbiota-targeted interventions could help to alleviate or prevent the distressing side-effects of antipsychotic medications. The investigators have previously published promising data demonstrating anti-obesity effects of a novel Bifidobacterium longum APC1472, in a mouse model of obesity and in an overweight/obese population of humans, reducing levels of glucose and normalizing ghrelin levels. Because atypical antipsychotic medications are often used in people experiencing psychosis and the mechanisms of antipsychotic-induced weight gain and metabolic dysfunction have been suggested to include glucose intolerance (hyperglycaemia) and aberrant ghrelin signalling, the investigators propose to assess if adjunct supplementation of Bifidobacterium longum APC1472 can attenuate weight gain and metabolic side-effects associated with the use of atypical antipsychotic medication in people with non- affective psychosis. The investigators propose an exploratory patient-oriented research study, to assess the potential of adjunct Bifidobacterium longum APC1472 supplementation in individuals with psychosis receiving antipsychotic treatment, to ameliorate the liability to gain weight and/or normalize metabolic disturbances. Findings from this study will support clinical decision-making, increasing patient choice, and increase medication adherence, which will ultimately improve health and quality of life, and overall wellbeing of individuals as they pass through normal life stages.

A high percentage of individuals experiencing affective or a non-affective psychotic episode are treated with second-generation antipsychotics. While effective, most are associated with a significant liability for weight gain and metabolic disorders, negatively impacting adherence, health and quality of life. This study will explore the potential of a metabolically beneficial Bifidobacterium longum APC1472 to attenuate weight gain and metabolic side-effects in individuals with a non-affective psychosis, treated with antipsychotics.

ELIGIBILITY:
Inclusion Criteria:

* 8.1 Inclusion Criteria To be considered eligible for enrolment into the study, subjects must;

  1. Aged between 18-65 years old including women of child-bearing age
  2. Having a diagnosis of affective or non-affective functional psychosis defined according to ICD-10 criteria for psychosis (codes F20-30 & F32.3)
  3. Patients who are able to and have given written informed consent
  4. Patients who are willing to provide blood samples
  5. Patients who are willing to provide saliva (cortisol) and faecal microbiome samples
  6. Considering the nature of the study participants, a broad spectrum of concomitant medication will be permissible. Psychotropic meds, including antidepressants, mood stabilisers (lithium, valproate, carbamazepine), hypnotics and benzodiazapines, will be allowed as to not limit recruitment of this type of study participant.

Exclusion Criteria:

1. Intravenous drug use
2. Diagnosis of substance dependence in the past 3 months
3. Pregnancy or planning a pregnancy
4. Antibiotic use in the past 30 days
5. Steroid use in the past 30 days
6. Use of anti-coagulants, anti-inflammatory drugs, over-the counter non-steroidal anti-inflammatories (NSAIDS) and analgesics. Subjects should have a wash-out period of 4 weeks.
7. Patients suffering from any clinically significant or unstable medical condition, including congestive heart failure, coeliac disease, or an immunodeficiency syndrome.
8. Pre or probiotic supplements within the past 30 days.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-05-16 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Bifidobacterium longum on weight gain | change from baseline to 4, 8,12 weeks (end of study) and 18 weeks (washout)
  Investigate if supplementation with Bifidobacterium longum APC1472 capsules can attenuate weight gain in male and female human patients with psychosis treated with antipsychotics (olanzapine, clozapine, risperidone, paliperidone, aripiprazole, cariprazine and quetiapine).
  Primary outcome is the comparative end-point body weight (kg) between the placebo and probiotic groups to determine the effect of supplementation on antipsychotic-induced weight gain.
Bifidobacterium longum on glucose levels. | change from baseline to 4, 8, 12 weeks (end of study) and 18 weeks (washout)
  Investigate if supplementation with Bifidobacterium longum APC1472 capsules can attenuate fasting levels of glucose in male and female human patients with psychosis treated with antipsychotics (olanzapine, clozapine, risperidone, paliperidone, aripiprazole, cariprazine and quetiapine).
  Primary outcome is the comparative fasted glucose levels (measured in mg/dL or mmol/L) between the placebo and probiotic groups to determine the effect of supplementation on antipsychotic-induced high glucose levels.

SECONDARY OUTCOMES:
Bifidobacterium longum on waist-to-hip ratio | change from baseline to 4, 8, 12 weeks (end of study) and 18 weeks (washout)
  • Effect of APC1472 on waist-to-hip ratio
Bifidobacterium longum on metabolic syndrome markers | change from baseline to 4, 8, 12 weeks(end of study) and 18 weeks (washout)
  Markers related to metabolic syndrome and cardiometabolic function analysed (Blood pressure, HbA1C, cholesterol, LDL, HDL, triglycerides Cholesterol), measured in mg/dL or mmol/L, pg/mL, (mmHg), mmol/mol or percent (%), where appropriate.
Bifidobacterium longum on cortisol awakening response | change from baseline to 4, 8, 12 weeks (end of study) and 18 weeks (washout)
  • Saliva samples assessed for cortisol awakening response (µg/dL or nmmol/L) and correlated with weight gain and metabolic markers.
Bifidobacterium longum on treatment adherence | change from baseline to 4, 8, 12 weeks (end of study) and 18 weeks (washout)
  Improvement in treatment adherence analysed using questionnaires (self-rated scales).
Bifidobacterium longum on changes in food intake behavior | change from baseline to 4,8, 12 weeks (end of study) and 18 weeks (washout)
  Changes in diet, appetite and food preference, using the FFQ and the Leeds Food Preference Questionnaire.

OTHER OUTCOMES:
Bifidobacterium longum on neuroendocrine signalling | change from baseline to 4, 8, 12 weeks (end of study) and 18 weeks (washout)
  • Exploratory outcomes measuring endocrine hormones, including ghrelin (active and total), leptin, insulin, PYY, GLP-1 (active and total) in pmol/L or pg/mL.
Bifidobacterium longum on inflammatory markers | change from baseline to 4, 8, 12 weeks (end of study) and 18 weeks (washout)
  • Exploratory outcomes measuring C-peptide (CRP), and other inflammatory cytokine levels (IFNγ, Il-4, IL-6 Il-10, TNF-a) in pmol/L or pg/mL.
Bifidobacterium longum on gut microbiota | change from baseline to 4, 8, 12 weeks (end of study) and 18 weeks (washout)
  Microbiota analysis using shotgun metagenomic analysis, to investigate the impact of Bifidobacterium longum APC1472 supplementation on the gut microbiota composition, diversity and volatility in human patients treated with antipsychotics. Analysis will use taxonomic and functional readouts, including alpha and beta diversity index.

CONTACTS AND LOCATIONS:
Overall Officials: Harriet Schellekens, PhD, Principal Investigator — University College Cork
Locations (2):
- Ireland (2):
  - EIST clinics at St Mary's Primary Care Centre, Gurraunabraher & St Michaels In-Patient unit in the Mercy., Cork
  - RISE Metabolic Monitoring Clinics, Cork

IPD SHARING:
Plan to Share IPD: No